CLINICAL TRIAL: NCT06599268
Title: Women in Pharmaceutical Executive Roles: Analyzing the Barriers and Enablers for Women Reaching Top Executive Positions in Pharmaceutical Companies and Pharmacies
Brief Title: Analyzing the Barriers and Enablers for Women Reaching Top Executive Positions in the Pharmaceutical Sector
Acronym: POWER-BE
Status: Completed | Type: Observational
Sponsor: Lebanese University (Other)
Responsible Party: Principal Investigator, Georges Hatem, Associate Researcher, Lebanese University
Other Study IDs: 17/24/D
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Perception, Self

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pharmacists: Pharmacists/Pharmacy Students working in pharmaceutical companies or communities among others
  Interventions: Behavioral: Survey using a questionnaire.

INTERVENTIONS:
Behavioral: Survey using a questionnaire. — Questionnaire to assess the barriers and enablers for women reaching top executive positions in pharmaceutical companies and pharmacies
  The following sections will be considered:
  * General Characteristics of the Participants
  * Work-related characteristics
  * Barriers faced by women to reach top executive positions (Likert scale)
  * Enablers for women to reach top executive positions (Likert scale)
  * Conception of women in the pharmaceutical sector (Likert scale)

SUMMARY:
Research into the barriers and enablers for women's advancement in the pharmaceutical sector highlights several key factors. On the one hand, systemic issues such as gender bias, the glass ceiling, and the lack of adequate mentorship prevent many women from reaching executive roles. These barriers are often compounded by societal expectations, family responsibilities, and the rigid structures of work environments that disproportionately affect women. On the other hand, enabling factors like strong mentorship, diversity policies, leadership development programs, and workplace flexibility have proven to help women overcome these challenges and climb the corporate ladder. Companies that actively promote inclusive cultures and provide opportunities for women to develop leadership skills have seen greater success in gender diversity at the executive level.

Understanding the dynamics of women's leadership in pharmaceuticals is particularly relevant in regions like Lebanon, where cultural and social norms heavily influence gender roles. Although women in Lebanon are increasingly pursuing careers in healthcare and pharmaceuticals, few reach executive positions due to a combination of cultural expectations and structural limitations within companies. Analyzing the barriers and enablers for women's leadership in this context is crucial, as Lebanon's healthcare and pharmaceutical sectors play a vital role in the country's economy and well-being. Including women in leadership roles could enhance decision-making, foster innovation, and lead to more balanced workplace environments. Moreover, in a country with a history of political instability and economic challenges, addressing gender disparity in leadership becomes not just a matter of equality but one of economic necessity. Women bring diverse perspectives and leadership styles that can help companies navigate complex markets, drive performance, and foster sustainability. In the Lebanese pharmaceutical sector, where the demand for skilled professionals and innovative leadership is high, unlocking the potential of women in executive roles can lead to more resilient and adaptable organizations.

DETAILED DESCRIPTION:
The study titled Women in Pharmaceutical Executive Roles: Analyzing the barriers and enablers for women reaching top executive positions in pharmaceutical companies and pharmacies; focuses on exploring the factors that either hinder or support women in attaining leadership positions in the pharmaceutical industry.

Overview:

Context: The pharmaceutical industry has a notable gender disparity in executive roles, despite significant female participation in the workforce. Women often face systemic barriers like gender bias, lack of mentorship, and societal expectations that limit their upward mobility.

Region of Focus: Lebanon, where cultural norms play a substantial role in shaping gender roles. Despite women being increasingly involved in healthcare, few reach executive positions due to these societal and structural barriers.

Objective: The study aims to identify these barriers and enablers to improve gender diversity in leadership, especially in Lebanon s pharmaceutical sector, which is crucial for its economy.

Methodology:

Population: The study targets pharmacists and pharmacy students working in pharmaceutical companies and pharmacies.

Exposure: It examines personal perceptions of workplace environments, especially in the context of Lebanon s post-pandemic and economic crisis.

Comparison and Data Collection: A questionnaire was designed to assess barriers and enablers using Likert scales across various sections:

General characteristics of participants Work-related characteristics Barriers faced by women in reaching executive roles Enablers for women's advancement Perceptions of women in the pharmaceutical sector Setting: The questionnaire is distributed online via platforms like Facebook, WhatsApp, and LinkedIn, aiming for 275 respondents. The data collection started in July 2024 and is ongoing.

Expected Outcomes:

Final theses for three MBA students at the Lebanese University, Faculty of Pharmacy.

A scientific publication in a peer-reviewed journal. A poster presentation at an international conference.

The study aims to highlight the importance of inclusive company cultures and leadership development programs that can pave the way for women to climb to executive positions in the pharmaceutical sector, ultimately fostering more innovative and adaptable organizations in Lebanon .

ELIGIBILITY:
Inclusion Criteria:

* Pharmacists/Pharmacy Students
* Working in companies/Community pharmacies

Exclusion Criteria:

* Non-Lebanese
* Those unemployed or Free-lancer
* Those working for companies outside Lebanon

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pharmacists/Pharmacy Students working in pharmaceutical companies
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation between the score of the schemes, as mentioned earlier, and the participants general characteristics. | through study completion, an average of 3 months
  The likert scale per scheme will be transformed into a score and associated with the participants characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Georges Hatem, Principal Investigator — Lebanese University
Locations (1):
- Lebanese University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided